CLINICAL TRIAL: NCT02084420
Title: PhaseⅢ Study of A Multicenter, Randomized, Double-blind, Active-controlled to Evaluate of Efficacy /Safety as H. Pylori Eradication Effect Between Ilaprazole/Pantoprazole
Brief Title: Efficacy/Safety Study as H. Pylori Eradication of Triple Therapy for 7 Days Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IY-81149-HB03
Record Dates: First submitted 2014-03-05; First posted 2014-03-12 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer | interventions — ilaprazole; Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ilaprazole or Pantoprazole placebo (Experimental): Ilaprazole 10mg, Pantoprazole 40mg, Amoxicillin 1000mg, Clarithromycin 500mg 2 times/day, PO
  Interventions: Drug: Ilaprazole
- Ilaprazole placebo or Pantoprazole (Active Comparator): Pantoprazole 40mg, Ilaprazole 10mg, Amoxicillin 1000mg, Clarithromycin 500mg 2 times/day,PO
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Ilaprazole — 10mg 2 BID( 2 times / day), before breakfast and dinner
  Other Names: NOLTEC
  Arms: Ilaprazole or Pantoprazole placebo
Drug: Pantoprazole — 40mg, BID(2 times / day), before breakfast and dinner
  Other Names: PANTOLOC
  Arms: Ilaprazole placebo or Pantoprazole

SUMMARY:
The purpose of this study is to evaluate of efficacy and safety as H.pylori eradiation effect between Ilaprazole and Pantoprazole triple therapy for 7 days treatment in Gastric and/or Duodenal ulcer patients with H.pylori positive infection.

DETAILED DESCRIPTION:
This study is to evaluate of efficacy and safety as H.pylori eradiation effect between Ilaprazole and Pantoprazole triple therapy for 7 days treatment in Gastric and/or Duodenal ulcer patients with H.pylori positive infection.

ELIGIBILITY:
Inclusion Criteria:

* 18 year old ≤ Male or female < 75 year old
* Patients who had endoscopically confirmed Gastric and/or duodenal ulcer and H.pylori infection confirmed by Urea Breath Test
* Patients who understand the study conditions
* Patients who had been given the explanation about the study, and had provided voluntary written informed consent to participate in the stud

Exclusion Criteria:

* Patients with known allergy or hypersensitivity reaction to the Investigational products
* Patients who use the Investigational products
* Patients who undergone H.pylori eradication
* Patients with abnormal laboratory results, as specified below:

Total bilirubin, creatinine > 1.5 x upper limit of normal Aspartate transminase, Alanine transminase, Alkaline phosphatase, Blood urea nitrogen > 2 x upper limit of normal

* Patients who used Proton Pump Inhibitor agents or antibiotics within the last 2 weeks before the start of the Investigational products
* Pregnant women and lactating women
* Women of childbearing potential who were not using a medically acceptable method of contraception during the study period.(Menopausal women who did not have a menstrual period for at least 12 months were considered infertile)
* Patients with uncontrolled Diabetes mellitus
* Patients with uncontrolled Hypertension
* Patients with Alcoholics
* Patients with a history of malignancy within 5 years prior to the study entry (Day 1) (except for basal cell carcinoma of the skin)
* Patients who had undergone a esophageal or gastric surgery
* Patients who had a hereditary disorder as galactose intolerance, lactose intolerance, glucose-galactose malabsorption
* Patients who had participated in other investigational study within 30 days before the study entry (Day 1)
* Patients who, in the investigator's opinion, are not suitable for the study for any other reason

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
the rate of H.pylori eradication | participants will be followed at 7 weeks (visit 4)

SECONDARY OUTCOMES:
the rate of Gastric and/or Duodenal ulcer curation | participants will be followed at 7 weeks (visit 4)

CONTACTS AND LOCATIONS:
Overall Officials: IL YANG PHARM, Study Director — IL-YANG Pharmaceutical Co.LTD
Locations (18):
- South Korea (18):
  - Soonchunhang University Hospital, Bucheon-si, Gyeonggi-do
  - Inje Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Gachon University Gill Medical Center, Incheon
  - Wonkwang University of Medicine & Hospital, Jeollabuk-do
  - Chung Ang University Hospital, Seoul
  - Ewha Womens University Mokdong Hospital, Seoul
  - Inje University Seoul Paik Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - KyungHee University Medical center, Seoul
  - Seoul Asan hoapital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul, Seoul
  - Wonju Severance Christian Hospital, Wonju-si, Gangwon-do